CLINICAL TRIAL: NCT04075604
Title: Randomized, Non-comparative Neoadjuvant Phase II Study in Patients With ER+/HER2- Breast Cancer >= 2 cm With Safety Run-in, Assessing Nivolumab + Palbociclib + Anastrozole
Brief Title: A Study of Neoadjuvant Nivolumab + Palbociclib + Anastrozole in Post-Menopausal Women and Men With Primary Breast Cancer
Acronym: CheckMate 7A8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7A8
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Cancer
Keywords: Nivolumab; Breast Cancer; Cancer; ER+; HER2-; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Nivolumab; Anastrozole; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Nivolumab+Palbociclib+Anastrozole (ANZ) (Experimental)
  Interventions: Biological: Nivolumab; Drug: Anastrozole; Drug: Palbociclib
- Arm B: Palbociclib+ANZ then Nivolumab+Palbociclib+ANZ (Experimental)
  Interventions: Biological: Nivolumab; Drug: Anastrozole; Drug: Palbociclib
- Arm C: Palbociclib+ANZ (Active Comparator)
  Interventions: Drug: Anastrozole; Drug: Palbociclib

INTERVENTIONS:
Biological: Nivolumab — Specified Dose on Specified Days
  Arms: Arm A: Nivolumab+Palbociclib+Anastrozole (ANZ); Arm B: Palbociclib+ANZ then Nivolumab+Palbociclib+ANZ
Drug: Anastrozole — Specified Dose on Specified Days
Drug: Palbociclib — Specified Dose on Specified Days

SUMMARY:
A randomized multi-arm study evaluating the safety and efficacy of palbociclib and anastrozole with or without nivolumab in participants with ER+/HER2- breast cancer

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Participants must have untreated, unilateral, histologically confirmed ER+, HER2- invasive breast cancer with primary tumor ≥2 cm in largest diameter (cT1-3) in one dimension by clinical or radiographic exam, for whom neoadjuvant endocrine monotherapy deemed to be a suitable therapy.
* Participants must be deemed eligible for surgery and must agree to undergo surgery after completion of neoadjuvant therapy and agree to provide tumor tissue at baseline, on-treatment, and at surgery.
* Women must have documented proof that they are not of childbearing potential.
* Participants must have a performance status (PS) ≤ 1 on the Eastern Cooperative Oncology Group (ECOG) scale

Exclusion Criteria:

* Participants who may have had any treatment, including radiotherapy, chemotherapy, and/or targeted therapy administered for the currently diagnosed breast cancer prior to enrollment or for whom upfront chemotherapy is clinically judged appropriate as optimal neoadjuvant treatment.
* Participants who have a history of or active, known or suspected autoimmune disease, or other syndrome that requires systemic steroids above physiological replacement dose or autoimmune agents for the past 2 years.
* Prior treatment with either ET or CDK4/6 inhibitors for Breast Cancer (BC) within 5 years or an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways, or history of allergy, or hypersensitivity to study drug components
* Prior malignancy active within the previous 3 years or participants with serious or uncontrolled medical disorders.
* Personal history of any of the following conditions: syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), long or short QT syndrome, Brugada syndrome, or known history of corrected QT prolongation, Torsade de Pointes, or sudden cardiac arrest.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (36):
- United States (9):
  - Local Institution - 0031, Whittier, California
  - University Cancer Blood Ctr, Athens, Georgia
  - Northside Hospital,Inc.- Central Research Department, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Local Institution - 0041, Florham Park, New Jersey
  - The Cancer Center At Hackensack University Medical Center, Hackensack, New Jersey
  - MetroHealth Medical Center, Cleveland, Ohio
  - Hematology-Oncology Associates Of Fredricksburg, Inc, Fredericksburg, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
- Australia (2):
  - Local Institution - 0005, Elizabeth Vale, South Australia
  - Breast Cancer Research Centre - WA, Nedlands, Western Australia
- Belgium (3):
  - Local Institution - 0011, Wilrijk, Antwerpen
  - Local Institution, Liège
  - Local Institution, Namur
- Local Institution - 0071, Ottawa, Ontario, Canada
- France (7):
  - Local Institution - 0075, Bordeaux
  - Local Institution - 0073, Créteil
  - Local Institution - 0072, La Roche-sur-Yon
  - Centre Leon Berard, Lyon
  - Local Institution - 0019, Marseille
  - Centre de Cancerologie du Grand Montpellier, Montpellier
  - Institut Claudius Regaud, Toulouse
- Germany (5):
  - Local Institution, Bonn
  - Local Institution, Erlangen
  - Klinik Essen-Mitte, Essen
  - Local Institution, Mönchengladbach
  - Local Institution, Saarbrücken
- Puerto Rico (3):
  - Local Institution - 0047, Monterrey Ponce
  - Local Institution - 0002, San Juan
  - Local Institution - 0062, San Juan
- Spain (6):
  - H. Univ. Vall dHebron, Barcelona
  - Local Institution - 0037, Barcelona
  - Hosp Univer 12 De Octubre, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario De Valencia, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Dose Level 1: Nivolumab: 480 mg every 4 weeks (Q4W) intravenously (IV) Abemaciclib: 150 mg twice daily (BID) per os (by mouth) Anastrozole: 1 mg once daily (QD) per os (by mouth) Participants will be treated for a maximum of 5 cycles (1 cycle = 4 weeks)
- Cohort 2: Dose Level 1: Nivolumab: 480 mg every 4 weeks (Q4W) intravenously (IV) Palbociclib: 125 mg once daily (QD) per os (by mouth) for 3 weeks of each cycle (1 week off) Anastrozole: 1 mg once daily (QD) per os (by mouth) Participants will be treated for a maximum of 5 cycles (1 cycle = 4 weeks)
- Cohort 2: Dose Level 2: Nivolumab: 480 mg every 4 weeks (Q4W) intravenously (IV) Palbociclib: 100 mg once daily (QD) per os (by mouth) for 3 weeks of each cycle (1 week off) Anastrozole: 1 mg once daily (QD) per os (by mouth) Participants will be treated for a maximum of 5 cycles (1 cycle = 4 weeks)
Period: Overall Study
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Started | 2 | 9 | 12
Completed | 1 | 3 | 6
Not Completed | 1 | 6 | 6
Not completed — Adverse Event | 0 | 0 | 3
Not completed — Participant request to discontinue study treatment | 0 | 0 | 1
Not completed — Participant withdrew consent | 0 | 0 | 1
Not completed — Other reasons | 1 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0
Not completed — Study drug toxicity | 0 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2 | Total
Number analyzed (Participants) | 2 | 9 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (2.8) | 60.3 (9.3) | 67.4 (10.2) | 64.3 (9.8)
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 1 | 7 | 5 | 13
  >= 65 AND < 75 | 1 | 1 | 3 | 5
  >= 75 AND < 85 | 0 | 1 | 4 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 12 | 23
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 2 | 5 | 7 | 14
  Unknown or Not Reported | 0 | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 9 | 11 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Dose Limiting Toxicities (DLT) in the Safety Run-in Phase
Description: The number of participants with dose limiting toxicities (DLTs) during the safety run-in phase. DLTS are defined as treatment emergent adverse events (TEAE) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 that occurs during the first 4 weeks (1 cycle) after treatment. Participants who withdraw from the study during the DLT evaluation period or have received less than 1 dose of nivolumab and 75% of accumulative doses of palbociclib of the cycle for reasons other than a DLT will not be considered as DLT-evaluable participants.
Time Frame: From first dose to 4 weeks after first dose
Population: All DLT-evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 1 | 9 | 12
Participants | 0 | 2 | 0

2. Primary Outcome: Residual Cancer Burden (RCB) 0-1 Rate in the Randomized Phase
Description: RCB 0-I rate is defined as the percentage of randomized participants who achieve RCB 0: no residual disease or RCB-I: minimal residual disease. RCB is a continuous index combining pathological measurements of primary tumor (size and cellularity) and nodal metastases (number and size) defined by a point system at surgery.
  No participants continued to the randomized phase; trial was closed after completion of the Safety Run-in.
Time Frame: From randomization phase up to 5 treatment cycles (up to approximately 20 weeks)
Population: All randomized participants in the Randomized phase.
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) per investigator radiographic assessment. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to approximately 6 months after first dose
Population: All Treated Participants in the Safety Run-in Phase
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Percentage of Participants | 0.0 [0.0 to 84.2] | 66.7 [29.9 to 92.5] | 75.0 [42.8 to 94.5]

4. Secondary Outcome: Breast Conserving Surgery (BCS) Rate
Description: The percentage of participants who undergo breast conserving surgery (BCS) after completing the study treatments. Confidence interval based on the Clopper and Pearson method.
Time Frame: From first dose up to approximately 6 months after first dose
Population: All Treated Participants in the Safety Run-In Phase
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Percentage of Participants | 50.0 [1.3 to 98.7] | 55.6 [21.2 to 86.3] | 50.0 [21.1 to 78.9]

5. Secondary Outcome: Pathological Complete Response (pCR) Rate
Description: The percentage of participants with an absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy. Confidence interval based on the Clopper and Pearson method.
Time Frame: From first dose up to approximately 6 months after first dose
Population: All Treated Participants in the Safety Run-In Phase
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Percentage of Participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 33.6] | 8.3 [0.2 to 38.5]

6. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: The number of participants experiencing adverse events (AEs). An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 6 months)
Population: All Treated Participants in the Safety Run-In Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants | 2 | 9 | 12

7. Secondary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: The number of participants experiencing serious adverse events (SAEs). A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 6 months)
Population: All Treated Participants in the Safety Run-In Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants | 0 | 5 | 2

8. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: The number of participants experiencing adverse events (AEs) that lead to discontinuation of study treatment. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 6 months)
Population: All Treated Participants in the Safety Run-In Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants | 0 | 5 | 4

9. Secondary Outcome: The Number of Participants Experiencing Immune-Related Adverse Events (AEs)
Description: The number of participants experiencing adverse events that are immune-related. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 8 months)
Population: All DLT-evaluable participants in the Safety Run-in Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 1 | 9 | 12
Participants
  Hypothyroidism | 1 | 0 | 0
  Hyperthyroidism | 0 | 0 | 1
  Immune-mediated lung disease | 0 | 1 | 0
  Pneumonitis | 0 | 0 | 1
  Hepatitis | 0 | 3 | 2
  Rash | 0 | 2 | 0

10. Secondary Outcome: The Number of Participants Deaths
Description: The number of participants that have died during the study.
Time Frame: From first dose up to approximately 8 months
Population: All Treated Participants in the Safety Run-In Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants | 0 | 0 | 0

11. Secondary Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Thyroid Tests - SI Units
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on SI conventional units.
  TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 6 months)
Population: All Treated Subjects in Safety Run-in Phase with at Least One On-Treatment TSH measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants
  TSH > ULN | 1 | 3 | 2
  TSH > ULN WITH TSH <= ULN AT BASELINE | 1 | 2 | 1
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 0 | 1 | 2
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0 | 2 | 2
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 0 | 0
  TSH < LLN | 0 | 3 | 4
  TSH <LLN WITH TSH >= LLN AT BASELINE | 0 | 2 | 4
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0 | 1 | 1
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0 | 1 | 3
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 1 | 0

12. Secondary Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Liver Tests
Description: The number of participants with laboratory abnormalities in specific liver tests based on SI conventional units.
  ALT = Alanine Aminotransferase AST = Aspartate Aminotransferase ULN = Upper Limit of Normal
Time Frame: From first dose to 30 days after last dose of study therapy (up to approximately 6 months)
Population: All Treated Participants in the Safety Run-in Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
Number analyzed (Participants) | 2 | 9 | 12
Participants
  ALT OR AST > 3XULN | 0 | 4 | 3
  ALT OR AST > 5XULN | 0 | 3 | 3
  ALT OR AST > 10XULN | 0 | 2 | 2
  ALT OR AST > 20XULN | 0 | 1 | 2
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 0
  ALP > 1.5XULN | 0 | 3 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 1 DAY | 0 | 1 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>1.5XULN IN 30 DAYS | 0 | 1 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were monitored from first dose to 100 days after last dose of study therapy (up to approximately 8 months). Serious Adverse events were monitored between first dose and 30 days after last dose of study therapy. (Up to approximately 6 months) Participants were assessed for All Cause Mortality from their first dose until the study was completed (up to approximately 21 months)
Arm/Group | Cohort 1: Dose Level 1 | Cohort 2: Dose Level 1 | Cohort 2: Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 5/9 | 3/12
Other Adverse Events (participants affected / at risk) | 2/2 | 8/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose Level 1 (N=2) | Cohort 2: Dose Level 1 (N=9) | Cohort 2: Dose Level 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dose Level 1 (N=2) | Cohort 2: Dose Level 1 (N=9) | Cohort 2: Dose Level 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 4
Axillary pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 5
Mucosal inflammation (General disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Xerosis (General disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 4 | 2
Amylase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 5
Platelet count decreased (Investigations) | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 2 | 2

LIMITATIONS AND CAVEATS:
Bristol Myers Squibb (BMS) decided to permanently discontinue enrollment and dosing in the nivolumab + abemaciclib + anastrozole cohorts during the Safety Run-in phase due to the risk of serious interstitial lung disease (ILD)/pneumonitis in patients receiving abemaciclib in combination with pembrolizumab. BMS decided to not move forward with the randomized phase of CA2097A8 and to close the trial after completion of the Safety Run-in.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT04075604/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04075604/SAP_001.pdf